CLINICAL TRIAL: NCT05239780
Title: Invasive Decoding and Stimulation of Altered Reward Computations in Depression
Brief Title: Invasive Decoding and Stimulation of Altered Reward Computations in Depression Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: University of California, Davis (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ignacio Saez, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-17-00258; 1R01MH124763-01 (NIH)
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-06

CONDITIONS: Major Depressive Disorder
Keywords: Electrophysiology; Stereotactic encephalography; Brain stimulation
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants with depression (Experimental): Participants with depression to undergo brain stimulation
  Interventions: Procedure: Brain stimulation

INTERVENTIONS:
Procedure: Brain stimulation — Brain stimulation will be performed after collection of clinical seizure data. Bipolar stimulation to one or several adjacent electrodes will be applied. Stimulation design will be either determined prior to testing or designed according to results from neurobehavioral assessments. Stimulation will consist of biphasic, constant-current trains of stimulation pulses at 100 Hz, with 100 ms pulse width or a sinusoidal wave of a predefined mean band frequency (i.e. 6Hz for θ, 11Hz for α, 20Hz for β, etc.). Stimulation intensity will be ≤6 mA, consistent with parameters used for clinical mapping, for the duration of the behavioral task or for short (2-3 s) periods of time at given epochs during the task (i.e. outcome evaluation). Clinical personnel will be available during stimulation to help monitor stimulation-induced after-discharges; if any are detected, stimulation intensity will be dialed down or terminated.

SUMMARY:
Novel invasive neurostimulation stimulation strategies through neurosurgical interventions are emerging as a promising therapeutical strategy for major depressive disorder. These have been applied mostly to the anterior cingulate cortex, but other limbic brain regions have shown promise as anatomical targets for new neurostimulation strategies. The researchers seek to study neural activity in limbic brain areas implicated in decision behavior and mood regulation to identify novel targets for treatment through electrical stimulation. To do this, the study team will record local field potentials (LFPs) from the orbitofrontal cortex, hippocampus and amygdala of epilepsy participants undergoing invasive monitoring (intracranial encephalography, iEEG) during choice behavior. Leveraging the high co-morbidity of depression and intractable epilepsy (33-50%), neural responses will be compared to reward across depression status to identify abnormal responses in depression. Finally, the researchers will use these as biomarkers to guide development of neurostimulation strategies for the treatment of depression.

DETAILED DESCRIPTION:
Participants (n=24) will complete a decision-making task in which participants will make decisions under uncertainty and seek to maximize rewards. The researchers will assess behavioral (risk attitudes) and neural (LFP) responses using a combination of intracranial recordings and computational modeling. A subset of patients will complete the game a second time under electrical stimulation of pre-identified anatomical targets in orbitofrontal cortex, hippocampus or amygdala. In addition, patients' depression status will be assessed through questionnaires (BDI-II and HDSA). Finally, the researchers will examine whether electrical stimulation results in behavioral or mood modulation.

ELIGIBILITY:
Inclusion Criteria:

- The study will follow clinical criteria for epilepsy patient recruitment for invasive monitoring. As a results, individuals of adults of all ages are expected to be included in this study.

Exclusion Criteria:

* Adults over 80 years of age will be excluded as per concerns of cognitive decline.
* Children under 18 will be excluded from the study since the maturation of frontal lobes continues through adolescence and significant differences in frontal lobe functioning between children younger than 18 and adults are often observed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Gambling Task | Day 1
  Risk attitudes will be evaluated behaviorally. Patients' behavior will in examined in experimental task (a gambling task) to determine overall proportion of risky choices (gambles) and indifference points (expected gamble value at which the patient is equally likely to choose a gamble or a safe bet). Score from 0%-100%, with higher percent indicating choosing the risky gamble more often.

SECONDARY OUTCOMES:
Beck's Depression I-II (BDI-II) score | Day 1
  Self-reported mood questionnaire. BDI-II total scale 0-63, with higher score indicating more severe depression.
Hamilton scales for depression and anxiety (HSDA) | Day 1
  HSDA comprise the Hamilton Depression Rating Scale (HDRS) and the Hamilton Anxiety Rating Scale (HAM-A). These are clinician-administered mood and anxiety reports. HDRS total score range from 0-81 with higher scores indicating greater depression severity. HAM-A total score range from 0-56, with higher score indicating higher severity. HRDS full scale from 0-137 where scores of 0-7 indicate normal range, whereas a score of 20 or higher indicates at least moderate severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Saez, Ph.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Any purpose. Proposals should be directed to ignacio.saez@mssm.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be included in the URL field below).